CLINICAL TRIAL: NCT07386600
Title: Perineural Dexamethasone Versus Perineural Dexmedetomidine as Adjuvants to Ropivacaine in iPACK and Adductor Canal Blocks for Total Knee Arthroplasty: A Randomized, Double-Blind, Controlled Trial
Brief Title: Dexamethasone vs Dexmedetomidine for iPACK + ACB in TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13/2025
Record Dates: First submitted 2025-12-04; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Patients receive ultrasound-guided iPACK block and adductor canal block (ACB) on the operative limb with ropivacaine 0.2% alone, without any perineural adjuvant.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Perineural Dexamethasone (Experimental): Patients receive ultrasound-guided iPACK and ACB with ropivacaine 0.2% combined with perineural dexamethasone.
  Interventions: Drug: Dexamethasone 4mg
- Perineural Dexmedetomidine (Experimental): Patients receive ultrasound-guided iPACK and ACB with ropivacaine 0.2% combined with perineural dexmedetomidine.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — Ultrasound-guided iPACK block and adductor canal block are performed using ropivacaine 0.2% in a standardized volume per block (20 mL for iPACK and 20 mL for ACB; adjust according to protocol). No adjuvant is added to the local anesthetic solution.
  Arms: Control
Drug: Dexamethasone 4mg — Ultrasound-guided iPACK block and adductor canal block are performed using ropivacaine 0.2% in a standardized volume per block (20 mL + 20 mL).
  Preservative-free dexamethasone is added to the local anesthetic solution at a dose of (2 x 2 mg).
  Arms: Perineural Dexamethasone
Drug: Dexmedetomidine — Ultrasound-guided iPACK block and adductor canal block are performed using ropivacaine 0.2% in a standardized volume per block (20 mL + 20 mL).
  Dexmedetomidine is added to the local anesthetic solution at a dose of 25ug, distributed between both blocks according to the study protocol
  Arms: Perineural Dexmedetomidine

SUMMARY:
This randomized, double-blind, controlled trial is designed to compare the analgesic efficacy and safety of perineural dexamethasone versus perineural dexmedetomidine as adjuvants to ropivacaine for ultrasound-guided interspace between the popliteal artery and the capsule of the posterior knee (iPACK) and adductor canal blocks in patients undergoing primary unilateral total knee arthroplasty (TKA). Elderly participants scheduled for elective TKA will be randomized into three parallel groups: ropivacaine alone (control), ropivacaine combined with perineural dexamethasone, or ropivacaine combined with perineural dexmedetomidine.

The primary objective is to determine whether the addition of either adjuvant reduces postoperative opioid consumption compared with ropivacaine alone and to assess potential differences in analgesic efficacy between the two adjuvants. Secondary outcomes include pain intensity at rest and during mobilization, time to first rescue analgesia, quality of early functional recovery, and the incidence of adverse events, including postoperative nausea and vomiting, motor impairment, and hemodynamic instability.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is associated with substantial postoperative pain, which may delay rehabilitation, prolong hospital stay, and increase opioid consumption. Ultrasound-guided peripheral nerve blocks are an integral component of multimodal analgesia for TKA, particularly the interspace between the popliteal artery and the capsule of the posterior knee (iPACK) block and the adductor canal block (ACB). These techniques provide effective analgesia while preserving quadriceps motor function, thereby facilitating early mobilization. Ropivacaine is the most commonly used local anesthetic for iPACK and ACB; however, its relatively limited duration often necessitates additional analgesic interventions.

Perineural adjuvants have attracted increasing interest as a means to prolong block duration and enhance the quality of peripheral nerve blockade. Dexamethasone and dexmedetomidine are among the most extensively studied adjuvants; however, their relative clinical efficacy and safety when administered perineurally in TKA remain uncertain. Dexamethasone has been shown to prolong block duration and reduce postoperative pain and opioid requirements, likely through anti-inflammatory and glucocorticoid-mediated mechanisms. Dexmedetomidine, an α2-adrenergic agonist, may further enhance analgesia and sensory block duration but has been associated with adverse effects such as sedation and bradycardia in susceptible patients. Comparative evidence between these agents in the specific context of combined iPACK and ACB is limited, and no clear consensus currently exists regarding their optimal use.

This randomized, double-blind, controlled clinical trial is designed to compare the efficacy and safety of perineural dexamethasone versus perineural dexmedetomidine as adjuvants to ropivacaine for ultrasound-guided iPACK and adductor canal blocks in elderly patients undergoing primary unilateral total knee arthroplasty. Eligible participants will be randomized into three parallel groups: ropivacaine alone (control), ropivacaine with perineural dexamethasone, or ropivacaine with perineural dexmedetomidine. All nerve blocks will be performed according to a standardized protocol by experienced anesthesiologists. Surgical, anesthetic, and postoperative analgesic management will be standardized across groups to minimize potential confounding factors. Participants, care providers, investigators, block practitioners, nursing staff, and outcome assessors will remain blinded to treatment allocation.

The primary outcome is cumulative opioid consumption during the first 24 postoperative hours, expressed as intravenous morphine equivalents. Secondary outcomes include pain intensity at rest and during mobilization, time to first rescue analgesia, motor-sparing profile, hemodynamic effects, quality of early recovery, and the incidence of adverse events such as postoperative nausea and vomiting, hypotension, bradycardia, and neurological symptoms. Functional recovery will additionally be evaluated using standardized physiotherapy milestones.

It is hypothesized that both perineural dexamethasone and dexmedetomidine will reduce postoperative opioid consumption compared with ropivacaine alone, and that one adjuvant may demonstrate superior analgesic efficacy or a more favorable safety profile. The findings of this study may provide clinically relevant evidence to guide the selection of perineural adjuvants for iPACK and adductor canal blocks in total knee arthroplasty, with the potential to improve pain control, accelerate rehabilitation, and reduce opioid exposure in an elderly, at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Scheduled for primary unilateral total knee arthroplasty under standardized anesthetic protocol
* ASA physical status II-III (or I-III, zależnie jak planujesz)
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Contraindications to peripheral nerve blocks (infection at injection site, coagulopathy, patient refusal)
* Known allergy or hypersensitivity to amide local anesthetics, dexamethasone or dexmedetomidine
* Chronic opioid therapy or opioid use > 30 mg oral morphine equivalents per day in the last 3 months
* Severe hepatic or renal impairment
* Significant cognitive impairment, inability to cooperate with pain assessment
* Participation in another interventional trial affecting pain or analgesic consumption

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours after surgery | 0-24 hours postoperatively
  Total dose of rescue opioid analgesics administered within the first 24 hours after surgery, converted to intravenous morphine equivalents (mg). All opioids given in the post-anesthesia care unit and on the ward will be recorded and converted using standard equianalgesic ratios.

SECONDARY OUTCOMES:
Pain intensity at rest | 6 hours postoperatively
  Pain intensity at rest assessed using an 11-point Numeric Rating Scale (NRS, 0 = no pain, 10 = worst imaginable pain)
Pain intensity at rest | 12 hours postoperatively
  Pain intensity at rest assessed using an 11-point Numeric Rating Scale (NRS, 0 = no pain, 10 = worst imaginable pain)
Pain intensity at rest | 24 hours postoperatively
  Pain intensity at rest assessed using an 11-point Numeric Rating Scale (NRS, 0 = no pain, 10 = worst imaginable pain)
Pain intensity at rest | 48 hours postoperatively
  Pain intensity at rest assessed using an 11-point Numeric Rating Scale (NRS, 0 = no pain, 10 = worst imaginable pain)
Pain intensity during mobilization | 24 hours postoperatively
  Pain during active knee flexion and mobilization (e.g., physiotherapy session) assessed using NRS (0-10)
Pain intensity during mobilization | 48 hours postoperatively
  Pain during active knee flexion and mobilization (e.g., physiotherapy session) assessed using NRS (0-10)
Time to first rescue analgesia | 0-48 hours postoperatively
  Time from completion of the iPACK and ACB blocks to the administration of the first dose of rescue opioid analgesic (in minutes).
Incidence of postoperative nausea and vomiting (PONV) | 0-48 hours postoperatively
  Number of patients with at least one episode of nausea and/or vomiting requiring antiemetic treatment during the first 24 and 48 hours after surgery.
Motor function of the operated limb | 6 hours postoperatively
  Quadriceps muscle strength (knee extension and hip adduction) assessed using the Medical Research Council (MRC) scale, ranging from 0 (no muscular contraction) to 5 (normal strength), to evaluate the motor-sparing profile of each analgesic regimen.
Motor function of the operated limb | 12 hours postoperatively
  Quadriceps muscle strength (knee extension and hip adduction) assessed using the Medical Research Council (MRC) scale, ranging from 0 (no muscular contraction) to 5 (normal strength), to evaluate the motor-sparing profile of each analgesic regimen.
Motor function of the operated limb | 24 hours postoperatively
  Quadriceps muscle strength (knee extension and hip adduction) assessed using the Medical Research Council (MRC) scale, ranging from 0 (no muscular contraction) to 5 (normal strength), to evaluate the motor-sparing profile of each analgesic regimen.
Block-related and systemic adverse events | Intraoperative and up to 48 hours postoperatively
  Incidence of bradycardia, hypotension, oversedation, local anesthetic systemic toxicity (LAST), neurological deficits, signs of infection at the injection site, or any serious adverse events possibly related to the study drugs or blocks.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, MD PhD, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the published article will be made available after de-identification. Data will include demographic characteristics, perioperative variables, intervention details, and primary and secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available beginning 6 months after publication of the main results and for a period of at least 5 years.
Access Criteria: Data will be shared with qualified researchers for legitimate scientific purposes upon reasonable request. Access requires submission of a methodologically sound proposal, approval by the study investigators, and a data use agreement.